CLINICAL TRIAL: NCT03595462
Title: The Benefits of Consuming Hummus as an Afternoon Snack on Appetite Control, Daily Food Intake, and Diet Quality in Adults
Brief Title: The Benefits of Consuming Hummus as an Afternoon Snack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Heather Leidy, Associate Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1804020480
Record Dates: First submitted 2018-06-30; First posted 2018-07-23 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior | interventions — Snacks

STUDY DESIGN:
Intervention Model Description: tightly-controlled, randomized cross-over design
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Snack (Experimental): The study participants will be provided with a snack to consume every day of the week. The energy content of the snacks will be standardized to ~240 kcal. The snacks will have different levels of protein, fat, carbohydrates, sugar, and fiber.
  Interventions: Other: Snack
- No Snack (Placebo Comparator): The study participants will not be provided with any snack and will be told to consume nothing from 2-4pm for a week.
  Interventions: Other: No Snack

INTERVENTIONS:
Other: Snack — Hummus and Pretzels- The study participants will be provided with a hummus and pretzels snack to consume every day for a week. The energy content of the hummus and pretzels will be ~240 kcal. The hummus and pretzels contain 6 g protein, 27 g carbohydrates, 0 g sugar, 4 g fiber, and 12 g fat.
  Granola Bars- The study participants will be provided with two granola bars to consume every day for a week. The energy content of the two granola bars will be ~240 kcal. The two granola bars contain 4 g protein, 38 g carbohydrates, 16 g sugar, 2 g fiber, and 9 g fat.
  Arms: Snack
Other: No Snack — The study participants will not be provided with any snack and will be told to consume nothing from 2-4pm for a week.
  Arms: No Snack

SUMMARY:
The investigators propose a randomized snack study in normal to overweight adults that will test whether the consumption of different afternoon snacks will have different effects on appetite, mood, blood sugar control, and food intake.

Aim 1: To examine whether the addition of hummus as part of an afternoon snack will improve diet quality, particularly through assessments of daily:

* Vegetable consumption
* Snacking behavior
* Energy intake
* Food choices

Aim 2: To examine whether the addition of hummus as part of an afternoon snack will improve appetite control and satiety including assessments of:

* Appetite Control (hunger, desire to eat, prospective food consumption)
* Cravings (sweet, salty, savory)
* Satiety (fullness)
* Eating initiation

Aim 3: To examine whether the addition of hummus as part of an afternoon snack will improve free-living glycemic control.

Aim 4: To explore whether the addition of hummus as part of an afternoon snack will improve mood/energy states

DETAILED DESCRIPTION:
Experimental Design: For 6 consecutive days/treatment, the participants will consume either hummus and pretzels, granola bars, or no snack between 2-4 pm and refrain from eating anything else during this time. On day 7, the participants will consume a standard breakfast, at home, and will come in to the investigator's facility 1 h prior to their habitual lunch time. The participants will be placed in a comfortable room, void of all time cues and a standardized lunch will be consumed. At 3 h after lunch, the participants will complete baseline appetite, satiety, and mood questionnaires. The respective snack will be given to the participants, and they will have 20 minutes to eat the snack. Snack palatability will also be assessed. The participants will continue to complete the previous questionnaires until they voluntarily choose to eat (again). At 3 h after snack, they will be presented with ad libitum dinner and evening snacks. They will be permitted to eat as much or as little as they would like to eat over the remainder of the day. In addition, from day 3 to day 8 of the testing week, continuous glucose monitoring will be completed to assess glucose control.

ELIGIBILITY:
Inclusion Criteria:

* normal to overweight (BMI: 18-32 kg/m2)
* no metabolic, psychological, or neurological diseases/conditions not currently or previously on a weight loss or other special diet (in the past 6 months)
* non-smoking
* not been clinically diagnosed with an eating disorder
* habitually eat an afternoon snack between 2:00-4:00 pm
* no food allergies related to the study snacks
* rates the overall liking of hummus higher than "Neither Like nor Dislike" on the screening palatability questionnaire.

Exclusion Criteria:

* Clinically diagnosed with an eating disorder
* Metabolic, hormonal, and/or neural conditions/diseases that influence metabolism or appetite
* Currently or previously on a weight loss or other special diet (in the past 6 months)
* Gained/lost >10 lb. over the past 6 months
* Taking medication that would directly influence appetite (weight-loss drugs or antidepressant, steroid, or thyroid medication, unless dosage has been stable for at least 6 months)
* Not willing or able to complete all study testing procedures

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Perceived Hunger | -180 min, -120 min, -60 min, +0 min, + 30 min, +60 min, +90 min, +120 min, +150 min, +180 min
  A questionnaire assessing perceived hunger will be completed at specific times throughout each of the the 6-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min) to 100 (max). A summation (area under the curve) will be calculated. Snacks were consumed at +0 min.
Perceived Fullness | -180 min, -120 min, -60 min, +0 min, + 30 min, +60 min, +90 min, +120 min, +150 min, +180 min
  A questionnaire assessing perceived fullness will be completed at specific times throughout each of the the 6-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min) to 100 (max). A summation (area under the curve) will be calculated. Snacks were consumed at +0 min.
Perceived Desire to Eat | -180 min, -120 min, -60 min, +0 min, + 30 min, +60 min, +90 min, +120 min, +150 min, +180 min
  A questionnaire assessing perceived desire to eat will be completed at specific times throughout each of the the 6-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min) to 100 (max). A summation (area under the curve) will be calculated. Snacks were consumed at +0 min.
Perceived Prospective Food Consumption | -180 min, -120 min, -60 min, +0 min, + 30 min, +60 min, +90 min, +120 min, +150 min, +180 min
  A questionnaire assessing how much food could be consumed will be completed at specific times throughout each of the the 6-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min) to 100 (max). A summation (area under the curve) will be calculated. Snacks were consumed at +0 min.

SECONDARY OUTCOMES:
Perceived Sweet | -180 min, -120 min, -60 min, +0 min, + 30 min, +60 min, +90 min, +120 min, +150 min, +180 min
  A questionnaire assessing perceived sweet cravings will be completed at specific times throughout each of the the 6-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min) to 100 (max). A summation (area under the curve) will be calculated. Snacks were consumed at +0 min.
Perceived Salty | -180 min, -120 min, -60 min, +0 min, + 30 min, +60 min, +90 min, +120 min, +150 min, +180 min
  A questionnaire assessing perceived salty cravings will be completed at specific times throughout each of the the 6-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min) to 100 (max). A summation (area under the curve) will be calculated. Snacks were consumed at +0 min.
Perceived Savory | -180 min, -120 min, -60 min, +0 min, + 30 min, +60 min, +90 min, +120 min, +150 min, +180 min
  A questionnaire assessing perceived savory cravings will be completed at specific times throughout each of the the 6-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min) to 100 (max). A summation (area under the curve) will be calculated. Snacks were consumed at +0 min.
Perceived Sleepiness | -180 min, -120 min, -60 min, +0 min, + 30 min, +60 min, +90 min, +120 min, +150 min, +180 min
  A questionnaire assessing perceived sleepiness will be completed at specific times throughout each of the the 6-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min) to 100 (max). A summation (area under the curve) will be calculated. Snacks were consumed at +0 min.
Perceived Energy | -180 min, -120 min, -60 min, +0 min, + 30 min, +60 min, +90 min, +120 min, +150 min, +180 min
  A questionnaire assessing perceived energy state will be completed at specific times throughout each of the the 6-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min) to 100 (max). A summation (area under the curve) will be calculated. Snacks were consumed at +0 min.
Perceived Alertness | -180 min, -120 min, -60 min, +0 min, + 30 min, +60 min, +90 min, +120 min, +150 min, +180 min
  A questionnaire assessing perceived alertness will be completed at specific times throughout each of the the 6-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min) to 100 (max). A summation (area under the curve) will be calculated. Snacks were consumed at +0 min.
Ad libitum Snack Pack-out | 3 testing days
  Free-living energy intake will be assessed on the in-clinic testing day of each treatment. When the participant leaves the testing facility, the participant will be provided with an excess of snacks to consume, ad libitum, throughout the remainder of the day. The quantity of food provided will be ~50% more than their estimated, weight-maintaining energy intake. All food items will be initially weighed and recorded. The participants will be instructed to return all uneaten foods as well as all wrappers and containers from consumed food. Any partially eaten, returned items will be weighed accordingly. The daily energy content will be assessed from these pack-outs.
Glucose Excursions Change | 6 days for each treatment
  Free-living, glucose measures will be performed for 7 consecutive days using Continuous Glucose Monitoring Device. The participants will report to our facility during one afternoon for insertion. A small area on the participant's abdomen will be cleaned and the tiny glucose sensor will be inserted just under the skin and held in place with Tegederm. The sensor measures glucose every 10sec and records an average glucose value every 5min for up to 144h.Calibration is performed by 4 finger sticks/d with a glucose analyzer.
Perceived Snack Palatability | 2 testing days that include snacks
  A questionnaires assessing how much the snack is liked will be completed at specific times throughout the 4-h testing days. The questionnaire contains a 100 mm VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The range is 0 mm (min) to 100 (max). A summation (area under the curve) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Leidy, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States